CLINICAL TRIAL: NCT02823444
Title: Non-Contrast Enhanced Peripheral Magnetic Resonance Angiography
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 50494
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2020-01

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication; Peripheral Vascular Disease
Keywords: Magnetic Resonance Imaging; Magnetic Resonance Angiography
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Peripheral Vascular Disease: Gender distribution will be approximately equal. The age range is 18-95, with increased prevalence in the elderly population.
  Interventions: Other: Magnetic Resonance Angiography
- Control: In the initial sequence optimization stage, healthy volunteers will also be recruited.
  Interventions: Other: Magnetic Resonance Angiography

INTERVENTIONS:
Other: Magnetic Resonance Angiography — Subjects who agree to participate in the study and provide written informed consent will undergo three station (abdomen/pelvis, thighs, and calves/feet) contrast and non-contrast enhanced magnetic resonance angiography of the lower extremities. Study visits may be split into two imaging sessions to decrease the time the participant is in the scanner if necessary. For image quality review, several participant may undergo only abdomen/pelvis imaging.
  Performance of the non-contrast magnetic resonance angiography requires placement of magnetic resonance imaging compatible electrocardiography leads on the patient's chest, so that the heart rate can be monitored and images can be obtained timed to each individual patient's heart beat. Electrocardiography monitoring/gating is performed routinely, and is not investigational.

SUMMARY:
To systematically develop, test, and refine peripheral vascular electrocardiography-gated fast spin echo magnetic resonance imaging for the accurate diagnosis of peripheral arterial disease without gadolinium contrast.

To test prospectively the accuracy of fast spin echo in peripheral arterial disease patients, compared with bolus-chase and time-resolved gadolinium enhanced magnetic resonance angiography. Additionally, as a substudy of this project, we will compare our fast spin echo approach with alternative non-contrast-enhanced magnetic resonance imaging methods such as time-of-flight and steady-state gradient echo imaging.

The overarching goals of our research are to develop and validate a peripheral magnetic resonance imaging technique that accurately depicts anatomy and disease without exposing patients to exogenous contrast material and its associated risks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known or suspected periphery arterial disease will be recruited.
* In the initial sequence optimization stage, healthy volunteers will also be recruited for magnetic resonance angiography

Exclusion Criteria:

* Patients with moderate to end stage renal disease (estimated glomerular filtration rate < 30 ml/min/1.73m2). These patients will not be recruited as they will be unlikely to undergo routine contrast enhanced magnetic resonance angiography due to the risk of developing Nephrogenic Systemic Fibrosis.
* Pregnant patients. Gadolinium chelates are a FDA Category C drug, and therefore should be avoided in pregnancy.
* Claustrophobic healthy volunteers or any subject who is unable to lie flat for 60 minutes.
* Glomerular filtration rate < 60ml/min/1.72m2 and coexisting history of pro inflammatory conditions such as recent surgery, sepsis or major infection, arterial or venous thrombosis.
* Any history of nephrogenic systemic fibrosis
* Unable/ unwilling to give informed consent
* Medical contra-indications to magnetic resonance imaging: e.g. pacemakers, implanted defibrillators, cochlear implants, aneurysm clips, and prior/ current metal workers. Patients will be screened with a safety questionnaire.
* Clinically unstable patients
* Patients with newly placed stents will be excluded until 8 weeks post placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population will be patients recruited from the University of Utah and Salt Lake City Veteran Affairs Medical Center. The intended gender distribution of the subjects will be approximately equal. There will be no gender based enrollment restrictions. The age range of the subjects is 18-95. No children will be recruited, as peripheral arterial disease is a disease of adulthood, with increased prevalence in the elderly population. There are no enrollment restrictions based upon race or ethnic origin. Patients with stents may be included.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-04; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Image Analysis | 2 years
  Image analysis of the non-contrast and contrast enhanced magnetic resonance angiography images from each patient will be performed by experienced readers. Each regional endpoints will be provided by each of the independent readers using non-contrast and contrast enhanced magnetic resonance angiography techniques. Each regional endpoint also will be provided by a consensus of the readers using all of the data from the magnetic resonance angiography techniques. Mixed model regression will be used to compare imaging methods in terms of overall image quality and reader confidence, with each endpoint analyzed separately and represented for each extremity as an average over readers.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Lee, MD, PhD, MBA, Principal Investigator — University of Utah; Lei Zhang, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No